CLINICAL TRIAL: NCT02649114
Title: Treatment of Eating Disorders With and Without Childhood Trauma: A Randomized Controlled Trial
Brief Title: Eating Disorders With and Without Childhood Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modum Bad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/836-1
Record Dates: First submitted 2015-09-08; First posted 2016-01-07 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Eating Disorders; Stress Disorders, Post-traumatic
MeSH Terms: conditions — Feeding and Eating Disorders; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-Behavioural Therapy (Active Comparator): This version of CBT is based on techniques employed in evidence-based approaches to a transdiagnostic sample. The programme includes; individualized formulation, taking into account different maintaining factors across cases (e.g., nutritional and/or emotional drivers for binging); agenda setting; homework; change in diet (particularly to improve carbohydrate intake); diary-keeping; exposure; behavioral experiments; cognitive restructuring; and surveys. The behavioral change is maintained as a focus, along with changes in mood and cognitions.
  Interventions: Behavioral: Cognitive-Behavioural Therapy
- Compassion-Focused Therapy (Experimental): There are four main treatment elements to the program. Two of these are linked to the experience of being a therapy group. This involves patients providing compassionate support to other group members.The third treatment element involves compassionate mind training which mainly focuses on activating the soothing system via imagery and related practical exercises.The final element of the program aims to help patients improve their ability to use their wider social network to access support.
  Interventions: Behavioral: Compassion-Focused Therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioural Therapy
  Arms: Cognitive-Behavioural Therapy
Behavioral: Compassion-Focused Therapy
  Arms: Compassion-Focused Therapy

SUMMARY:
The combination of EDs (ED) and post-traumatic sequelae of childhood trauma leads to significant impairment, suffering and represents a public health concern because it is frequently associated with role impairment, and is frequently under-treated. Considering the severity of these conditions, there is a need to develop more effective treatments that are tailored to the specific needs of these patients as no conclusion has been made about the treatment of choice. To improve treatment it is critically important to study treatment effects and the mechanism of these effects.

DETAILED DESCRIPTION:
The overall aim of the current project is; (1) To build knowledge on how to best treat patients with ED with and without childhood trauma, (2) To develop our understanding about how change happens for these patients. The investigators will do this by compare two treatment models; (1) Compassion-Focused Therapy (CFT) and (2) Cognitive Behavioural Therapy (CBT), for EDs both treatment types delivered at Modum Bad Psychiatric Center, department of ED.

Patients included in this randomized controlled trial will receive treatment at Modum Bad, satisfy DSM-V criteria for ED and half of the patients will in addition have a history of childhood trauma. A total of 86 patients who have received either CFT or CBT are followed up two year after completion of the treatment. The study utilises a rich data set collected outcome measures at altogether 5 time points and process and sub-outcome measures at 13 time points. The investigators will take advantage of our established collaborative networks, both nationally and internationally and existing procedures, where all patients are assessed with the same clinical instruments based on current state-of-the-art methods.

ELIGIBILITY:
Inclusion Criteria:

* satisfying DSM-V criteria for ED and for half of the patients in addition
* have a history of childhood trauma.

Exclusion Criteria:

* current suicidal risk
* current psychosis
* ongoing trauma (e.g. current involvement in an abusive relationship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-08; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Global index from Eating Disorder Examination questionnaire | Pre, weekly during treatment, post, 12-months followup, through study completion, an average of 1 year
  Change from baseline in eating disorder symptoms on the dimensional scales on the Eating Disorder Examination questionnaire

SECONDARY OUTCOMES:
Symptom checklist 90 revised | Time Frame: pre, post and 12-months followup, through study completion, an average of 1 year
  Change from baseline to 12-months follow-up
Inventory of interpersonal problems | Pre, post and 12-months followup, through study completion, an average of 1 year
  Change from baseline to 12-months follow-up
Dissociative experiences scale II | Pretreatment, posttreatment and 12-months followup, through study completion, an average of 1 year
  Change from baseline to 12-months follow-up
Short form 36 | Pretreatment, posttreatment and 12-months followup, through study completion, an average of 1 year
  Change from baseline to 12-months follow-up
Self-compassion scale | Pretreatment, posttreatment and 12-months followup, through study completion, an average of 1 year
  Change from baseline to 12-months follow-up
Symptom checklist-5 | Pretreatment, weekly during treatment, posttreatment and 12-months followupthrough study completion, an average of 1 year
  Change from baseline to 12-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: KariAnne Vrabel, PhD, Principal Investigator — Modum Bad
Locations (1):
- Modum Bad, Vikersund, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eielsen HP, Vrabel K, Olofsson ME. <<Scaringly Safe>>: Therapeutic Processes in Longstanding Eating Disorders With Comorbid Avoidant Personality Disorders in the Recovered Case of Jade. J Clin Psychol. 2025 Aug;81(8):694-705. doi: 10.1002/jclp.23805. Epub 2025 Apr 23. PMID 40267178
- [Derived] Kopland MCG, Vrabel K, Melsom L, Hoffart A, Johnson SU. Self-compassion in eating disorders and childhood trauma: A study of within-person effects in a randomized controlled trial. Psychother Res. 2023 Jun;33(5):640-653. doi: 10.1080/10503307.2022.2149363. Epub 2023 Jan 11. PMID 36630619
- [Derived] Vrabel KR, Wampold B, Quintana DS, Goss K, Waller G, Hoffart A. The Modum-ED Trial Protocol: Comparing Compassion-Focused Therapy and Cognitive-Behavioral Therapy in Treatment of Eating Disorders With and Without Childhood Trauma: Protocol of a Randomized Trial. Front Psychol. 2019 Jul 18;10:1638. doi: 10.3389/fpsyg.2019.01638. eCollection 2019. PMID 31379673
- [Derived] Olofsson ME, Oddli HW, Hoffart A, Eielsen HP, Vrabel KR. Change processes related to long-term outcomes in eating disorders with childhood trauma: An explorative qualitative study. J Couns Psychol. 2020 Jan;67(1):51-65. doi: 10.1037/cou0000375. Epub 2019 Aug 1. PMID 31368720